CLINICAL TRIAL: NCT06116383
Title: Evaluation of Renal Perfusion With NIRS in Adult Patients Undergoing Laparoscopic Cholecystectomy.
Brief Title: Evaluation of Renal Perfusion With NIRS in Laparoscopic Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Savas Altinsoy, Associate Professor MD, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: NIRS
Record Dates: First submitted 2023-09-28; First posted 2023-11-03 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Pneumoperitoneum; Renal Injury
Keywords: laparoscopy; NIRS; N-GAL
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing laparoscopic cholecystectomy.: Basal rSO2 values will be recorded by placing NIRS probes under the 10-11th intercostal space in the bilateral posterior lateral flank region. Age, gender, BMI, ASA scores, Hb/Htc values, intraoperative hemodynamic parameters, NIRS values, N-GAL (preoperative, 2nd hour and 24th hour), urea/creatinine (preoperative, postoperative 24th hour) values of the patients will be recorded. .
  Interventions: Device: NIRS

INTERVENTIONS:
Device: NIRS — Renal perfusion will be evaluated with NIRS

SUMMARY:
The investigators aimed to show the renal damage caused by increased intra-abdominal pressure in laparoscopic surgeries and to investigate whether its reflection on NIRS would be clinically effective.The main question it aims to answer are:

Does pneumoperitoneum cause renal damage?

NRS monitoring will be performed in patients undergoing laparoscopic surgery. Preoperative and postoperative blood tests will be performed at certain hours. N-GAL, urea and creatinine values will be recorded.

DETAILED DESCRIPTION:
Renal NIRS monitoring will be performed in patients undergoing laparoscopic cholecystectomy surgery. Age, gender, BMI, ASA scores, hemogblin/hematocrit values, intraoperative hemodynamic parameters, NIRS values, N-GAL (preoperative, 2nd hour and 24th hour), urea/creatinine (preoperative, postoperative 24th hour) values of the patients will be recorded. .

Before the general anesthesia is performed, the renal tissues of the patients will be visualized by ultrasound, the skin-renal cortex distances will be measured, and suitable patients will be included in the study. Basal rSO2 values will be recorded by placing NIRS probes under the 10-11. intercostal space in the bilateral posterior lateral flank region.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergoing elective laparoscopic cholecystectomi surgery lasting longer than 60 minutes
* BMI:18-25
* skin-renal cortex distance measured less than 4 cm on ultrasound
* ASA I-III

Exclusion Criteria:

* patient who did not give consent
* patient who had renal operation before,
* infection, abscess, catheter in the perirenal region
* hemodynamically unstable patients,
* patients with renal pathology and abnormal kidney function tests,
* emergency cases

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergoing elective laparoscopic cholecystectomi surgery
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2023-11-10 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of renal damage caused by pneumoperitoneum with N-GAL by blood test | During laparoscopic cholecystectomy operation and within 24 hours postoperative
  Taking a blood test to evaluation N-GAL
Evaluation of renal damage caused by pneumoperitoneum with urea/creatinin by blood test | During laparoscopic cholecystectomy operation and within 24 hours postoperative
  Taking a blood test to evaluation urea/creatinine values

CONTACTS AND LOCATIONS:
Overall Officials: Savaş Altınsoy, MD, Study Chair — Ankara Etlik City Hospital
Locations (1):
- Department of Anesthesiology and Reanimation, University of Health Sciences, Diskapi Yıldırım Beyazit Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caliskan E, Sanal Bas S, Onay M, Kilic Y, Kayhan Erdogan G, Tokar B. Evaluation of renal oxygenization in laparoscopic pediatric surgery by near infrared spectroscopy. Pediatr Surg Int. 2020 Sep;36(9):1077-1086. doi: 10.1007/s00383-020-04709-w. Epub 2020 Jul 10. PMID 32651617